CLINICAL TRIAL: NCT06747897
Title: Retrospective Consumer Experience on Former Use of DIPROBASE Advanced Eczema Cream® UI 1613882
Brief Title: An Observational Study to Gather Real-World User Feedback on DIPROBASE® Advanced Eczema Cream in Adults and Children With Eczema or Dry Skin
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22924
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dermatitis, Atopic
Keywords: Dry skin / Xerosis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult users: Use of product 3 months prior to recruitment
  Interventions: Device: MINERAL OIL + PETROLATUM (DIPROBASE® Advanced Eczema Cream, BAY987534, UI 1613882)
- Caregivers of children (2-12 years old): Use of product 3 months prior to recruitment
  Interventions: Device: MINERAL OIL + PETROLATUM (DIPROBASE® Advanced Eczema Cream, BAY987534, UI 1613882)
- Caregivers of children (<2 years old): Use of product 3 months prior to recruitment
  Interventions: Device: MINERAL OIL + PETROLATUM (DIPROBASE® Advanced Eczema Cream, BAY987534, UI 1613882)

INTERVENTIONS:
Device: MINERAL OIL + PETROLATUM (DIPROBASE® Advanced Eczema Cream, BAY987534, UI 1613882) — Product experience is assessed based on the answers provided by participants on the questions provided to them using an online questionnaire.

SUMMARY:
This is an observational study which means only data are collected from participants about their experience and symptoms, who received their usual treatment without any intervention from the study sponsor.

Atopic dermatitis, also known as eczema, is a long-lasting skin disease that causes redness, swelling, dryness, cracking, and intense itching. Xerosis is the scientific wording to describe dry skin. This condition is caused by a weakened skin barrier that does not hold moisture well.

DIPROBASE® advanced eczema cream is already available for use in the UK. It moisturizes and protects the skin.

This study is being done to understand how people use DIPROBASE® Advanced Eczema Cream and how consistently they adhere to its recommended use in their daily routines. In this study, participants will be asked to fill in an online questionnaire about their eczema symptoms and experience with DIPROBASE® Advanced Eczema Cream.

No treatment advice will be given as a part of this study.

The main purpose of this study is to gather feedback from people in the UK who have used DIPROBASE® Advanced Eczema Cream to treat their eczema or their dry skin condition. To do this, researchers will collect the following information from participants:

* intensity of eczema symptoms
* whether the cream provides a cooling or soothing effect
* whether the cream helps to ease the symptoms like itchiness, pain, or dryness

It is planned to identify and collect user data from November 2024 to January 2025. Participants will be recruited through a consumer database available with an external partner or via social media.

In this study, only data are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Biological sex: M/F.
* Age: > or equal to 18 years of age.
* Mothers, fathers, grandparents, and other caregivers aged 18 years of age and above, who will report data on themselves, their children from 2 to 12 years of age or their infants under 2 years of age.
* Able to read and understand the language of the online questionnaire.
* Have used the product within the previous three (3) months.
* Agree that the data collected can be used for research, marketing and regulatory purposes.

Exclusion Criteria:

* Due to the real-world nature of the study, there are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focusses on two key populations:
  * Adult Population: Adults aged 18 years and above who have used DIPROBASE® Advanced Eczema Cream for their eczema management.
  * Pediatric Caregiver population: Adult caregivers of children aged 2-12 years and infants 2 years and under who have applied the product to treat their children/ward's eczema.
  Subjects will be recruited via a consumer panel / consumer database available with the external partner (contract research organization) and/or social media.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Overall intensity of the symptoms | Retrospective analysis over three months
  Subjects will be asked to complete an online questionnaire assessing the overall intensity of their symptoms over the past three months, using a 4-point scale (0-no symptoms to 4-severe symptoms).
Coolness or soothing effect | Retrospective analysis over three months
  Subjects will be asked to complete an online questionnaire assessing their experience with the product over the past three months, using a 7-point scale (0-strongly disagree to 7-strongly agree).
Symptoms relief (skin irritation, pain, dryness) | Retrospective analysis over three months
  Subjects will be asked to complete an online questionnaire assessing their experience with the product over the past three months, using a 7-point scale (0-strongly disagree to 7-strongly agree).

SECONDARY OUTCOMES:
Descriptive summary of product usage: frequency, reasons, and ease of use | Retrospective analysis over three months
  Subjects will be asked to complete an online questionnaire assessing various points on product utilization and product characteristics, i.e. the frequency with which they apply the product (once, twice, more than twice), the reasons for its use, whether they sought medical advice prior to commencing use, the number of consecutive days they used it, and their assessment of the ease of application (very easy, easy, neutral, difficult, very difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- IQVIA Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here for access to information about Bayer's transparency standards and Bayer studies. — http://clinicaltrials.bayer.com/